CLINICAL TRIAL: NCT02013479
Title: The Chronic Autoimmune Thyroiditis Quality Of Life Selenium Trial
Brief Title: Selenium Supplementation in Autoimmune Thyroiditis
Acronym: CATALYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steen Bonnema (Other)
Collaborators: Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Pharma Nord (Industry); The Danish Medical Research Council (Other); Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Steen Bonnema, Chief Physician, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK-CATALYST
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Autoimmune Thyroiditis
MeSH Terms: conditions — Thyroiditis, Autoimmune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SelenoPRECISE (Experimental): SelenoPRECISE
  Interventions: Dietary Supplement: SelenoPRECISE
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SelenoPRECISE — Produced by Pharma Nord ApS, Vejle, Denmark
  Arms: SelenoPRECISE
Dietary Supplement: Placebo — Produced by Pharma Nord ApS, Vejle, Denmark
  Arms: Placebo

SUMMARY:
Our aim is to investigate if selenium supplementation versus placebo adjuvant to the standard treatment with levothyroxine (LT4) in patients with autoimmune thyroiditis will lead to improved thyroid specific quality of life, and reduced autoimmune activity. The trial will include 472 participants (2 X 236) from four clinical trial sites.

DETAILED DESCRIPTION:
Background: Chronic autoimmune thyroiditis (AIT) is a common autoimmune disease that often leads to impaired function of the thyroid gland, increases in incidence with age, and has an 8-9 time female preponderance. Quality of life is often impaired and complaints persist in a considerable number of patients, even after restoration of euthyroidism. The autoimmune component of the disease has been suggested as an explanation for this. Selenium is a micro nutritive essential for human health and the thyroid gland has the highest selenium concentration of all human tissues. Selenoproteins catalyse thyroid hormone metabolism and anti-oxidative processes in thyrocytes. In addition they are important to immune function. In Denmark, patients with AIT have lower blood selenium concentration than the background population. The majority of 13 randomised trials have shown that selenium supplementation decreases serum thyroid peroxidase antibody levels (TPO-Ab) in patients with AIT, when compared with placebo. We hypothesise that adjuvant selenium may be beneficial in the treatment of AIT.

Objectives: To investigate if selenium supplementation versus placebo adjuvant to the standard treatment with levothyroxine (LT4) in patients with AIT will lead to improved thyroid specific quality of life, and reduced autoimmune activity.

Design and trial size: The CATALYST trial is an investigator-initiated randomised, blinded, multicentre clinical trial of selenium supplementation versus placebo in patients with AIT. The trial will include 472 participants (2 X 236) from four clinical trial sites.

Intervention and duration: The experimental intervention group will receive 200 μg selenium-enriched yeast as two oral tablets once daily for 12 months. The control group will receive two placebo tablets, identical in appearance, taste and smell, once daily for 12 months. Six months additional follow-up leads to a trial duration of 18 months. The experimental supplement will be SelenoPrecise® by Pharma Nord ApS.

Time schedule: July 2012 - February 2014: preparation, approval and trial registration . March 2014: first participant first visit. March 2016: last participant first visit. September 2017: last participant last visit. Autumn 2017: analysis of biological samples and data, preparation of manuscripts.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Serum-TPO-Ab ≥ 100 IU/mL measured within the last 12 months.
3. Receiving LT4 treatment.

   - Serum-TSH ≥ 4.0 mU/L measured prior to treatment initiation
4. Written informed consent.

Exclusion Criteria:

1. Previous diagnosis of toxic nodular goitre, Graves' hyperthyroidism, post-partum thyroiditis or thyroid associated orbitopathy (TAO).
2. Previous radioiodine therapy, anti-thyroid treatment or thyroid surgery.
3. Previous diagnosis of non-melanoma skin cancer.
4. Morbidity, rendering the participant unable to process patient reported outcomes or receive intervention during the trial.
5. Systemic immunomodulatory medication.
6. Other medication known to affect thyroid function.
7. Pregnancy, breastfeeding, or planned pregnancy within 18 months.
8. Allergy towards the components in the selenium or placebo pills.
9. Intake of selenium supplementation ≥ 55 μg/d.
10. Unable to read or understand Danish.
11. Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2014-06; Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Thyroid related quality of life | 12 months after initation of intervention
  Measured in composite score based on the ThyPRO questionnaire

SECONDARY OUTCOMES:
Thyroid peroxidase antibody concentration (TPO-Ab) | 12 months after initation of intervention
Levothyroxine (LT4) dosage | 12 months after initation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Steen J Bonnema, MD, DMSc, Principal Investigator — Odense University Hospital; Laszlo Hegedüs, MD, DMSc, Principal Investigator — Odense University Hospital; Kristian H Winther, MD, Principal Investigator — Odense University Hospital; Torquil Watt, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Per Cramon, MD, Principal Investigator — Rigshospitalet, Denmark; Ulla Feldt-Rasmussen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Åse K Rasmussen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Jeppe Gram, MD, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark; Nils J Knudsen, MD, DMSc, Principal Investigator — Bispebjerg Hospital, Denmark
Locations (4):
- Denmark (4):
  - Clinic of Medical Endocrinology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Endocrinology and Gastroenterology, Bispebjerg Hospital, Copenhagen
  - Department of Internal Medicine, Hospital of South West Denmark, Esbjerg
  - Department of Endorcrinology and Metabolism, Odense University Hospital, Odense

REFERENCES:
- [Derived] Larsen C, Winther KH, Cramon PK, Rasmussen AK, Feldt-Rasmusssen U, Knudsen NJ, Bjorner JB, Schomburg L, Demircan K, Chillon TS, Gram J, Hansen SG, Brandt F, Nygaard B, Watt T, Hegedus L, Bonnema SJ. Selenium supplementation and placebo are equally effective in improving quality of life in patients with hypothyroidism. Eur Thyroid J. 2024 Jan 1;13(1):e230175. doi: 10.1530/ETJ-23-0175. Online ahead of print. PMID 38215286
- [Derived] Winther KH, Watt T, Bjorner JB, Cramon P, Feldt-Rasmussen U, Gluud C, Gram J, Groenvold M, Hegedus L, Knudsen N, Rasmussen AK, Bonnema SJ. The chronic autoimmune thyroiditis quality of life selenium trial (CATALYST): study protocol for a randomized controlled trial. Trials. 2014 Apr 9;15:115. doi: 10.1186/1745-6215-15-115. PMID 24716668